CLINICAL TRIAL: NCT04114188
Title: Tacrolimus After rATG and Infliximab Induction Immunosuppression (RIMINI)
Acronym: RIMINI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Petra Reinke (Other)
Collaborators: Institut Klinické a Experimentální Medicíny (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. Petra Reinke, Prof. Dr. Petra Reinke, sponsor representative, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIMINI
Record Dates: First submitted 2018-10-15; First posted 2019-10-03 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Renal Transplant Rejection
Keywords: transplant medicine
MeSH Terms: interventions — Antilymphocyte Serum; Infliximab; Tacrolimus; Prednisolone

STUDY DESIGN:
Intervention Model Description: This is a confidence-interval-estimation based early phase design, aiming to estimate a plausible range of the population treatment effect which is not bound to a formal hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antithymocyte Immunoglobulin (Rabbit) (Experimental): rATG induction on day 0 & 1 post op
  Interventions: Drug: Antithymocyte Immunoglobulin (Rabbit)

INTERVENTIONS:
Drug: Antithymocyte Immunoglobulin (Rabbit) — 1st kidney transplant recipients (low risk: PRA/cPRA < 20%, no DSA) will receive short rATG induction (2x1.5 mg/kg) given perioperatively and on first postoperative day. All patients will receive one shot Infliximab mAb at day 2. Since POD1, maintenance IS consists of Tac and tapered steroids therapy.
  Other Names: Infliximab; Tacrolimus; Prednisolone

SUMMARY:
International multicenter open-label single-arm confidence-interval-estimation based Phase II clinical trial, aiming to estimate a plausible range of the proportion of patients experiencing efficacy failure in the population, to provide evidence for efficacy and safety of the induction regimen with rATG and infliximab and a go/no go rule for further clinical development.

DETAILED DESCRIPTION:
A total of 75 patients will receive the proposed induction regimen, with expected 68 completers accounting for drop-outs and non-compliances with the protocol. If up to 27 out of the 68 completers experience efficacy failure, a progression into a larger trial will be considered justifiable. If the number of patients experiencing efficacy failure is between 28 and 34 out of 68, the merits of a larger non-inferiority design will be considered depending on the risk/benefit assessment. If more than 34 out of the 68 completers experience efficacy failure, a progression into a larger trial would be considered unjustifiable. 1st kidney transplant recipients (low risk: PRA/cPRA < 20%, no DSA) will receive short rATG induction (2x1.5 mg/kg) given perioperatively and on first postoperative day. All patients will receive one shot Infliximab mAb at day 2. Since POD1, maintenance IS consists of Tac and tapered steroids therapy. All patients will be followed up for one year.

At the POD 0 the first rATG dose (1.5mg/kg) will be given according to the local practice and Methyprednisolon 500mg will be given before reperfusion. At the POD 1 patients will receive methylprednisolon 500mg i.v. followed by second rATG dose (1.5mg/kg). Infliximab 5mg/kg b.w. will be given in slow infusion on POD2. Tacrolimus will be given the first dose before surgery at dose 0.1 mg/kg and next from POD1 at 0.2mg/kg/day and doses adjusted according to blood trough levels (10-15 ng/mL, POD1-POD13, 5-8ng/mL POD 14-90, 4-6ng/mL POD >90. Prednison (or appropriate dose of methylprednisolone) will be initiated POD 2 at a dose of 20mg/day and slowly tapered down to 5 mg at the POD 7 (POD2: 20mg, POD3: 15mg, POD4-5: 10mg, POD6-7: 7,5mg, > POD7: 5mg).

ELIGIBILITY:
Inclusion Criteria:

1. Primary deceased-donor or living-donor kidney transplantation XML File Identifier: CJub4EkHas0e/mXDp2mGyZzEe9E= Page 22/33
2. Men and women (recipient) age >18 years and <70 years
3. Panel reactive antibody frequency/ calculated panel reactive antibody frequency (peak PRA/cPRA) <20%
4. Written informed consent
5. Diagnosis of end stage renal disease
6. Women of Childbearing Potential (WOCBP) must be using a highly effective method of contraception (Pearl-Index < 1) to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL]. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of clinical trial. Male participants with pregnant or nonpregnant WOCBP partner must use condoms.

Exclusion Criteria:

1. Previous transplantation
2. Combined kidney transplantation with other organ
3. Subjects receiving an allograft from a donor older than 65 years with elevated serum creatinine levels and/or treated diabetes.
4. Immunosuppressive therapy up to 6 months before transplantation
5. Planned induction therapy with depletion agents
6. EBV seronegativity
7. HIV positivity
8. Leukopenia < 3000 cells per microliter, thrombocytopenia < 100 000 cells per microliter
9. Biological therapy history with ATG, OKT3, anti TNF agents
10. Tuberculosis history
11. Cancer history (skin non-melanoma cancer excluded)
12. Anti HCV positivity, HBsAg positivity or HBV DNA positivity
13. Detectable donor specific antibodies (DSA) by solid phase assay (Luminex®)
14. Subjects with a known hypersensibility to any of the drugs used in this protocol
15. Subjects who have used any investigational drug within 30 days prior to enrolment in this clinical trial
16. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period, women who are pregnant or breastfeeding or women with a positive pregnancy test on enrolment
17. Subjects who are legally detained in an official institution
18. All contraindications against study medication (including auxiliary substances)
19. Interactions with study medication
20. Current treatment with one of the following substances:

    cyclosporine, tacrolimus, mycophenolate mofetil, azathioprine, rituximab, prednisone
21. Patients unwilling to consent to saving and propagation of pseudonymized medical data and/or biological samples for study reasons
22. Chronic heart failure (NYHA III, IV) at transplantation
23. Participation in other clinical trials (pharmaceutical trials)
24. persons dependent of the sponsor, investigator or investigative site
25. positive Quantiferon test (for TBC)
26. live vaccine treatment 30 days prior to enrolment in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of efficacy failure [(treated biopsy-proven acute rejection, graft loss, death, or loss to follow-up) and renal function (estimated glomerular filtration rate)] of the induction regimen | 12 months post transplantation
  Composite endpoint of efficacy failure of the induction regimen defined as occurrence of any of the following individual outcomes up to 12 months post transplantation (start of follow up at transplantation): acute rejection, graft loss or poor graft function defined as eGFR<40 ml/min.

SECONDARY OUTCOMES:
Prevalence of biomarker signatures at 6, 12 months of follow-up. | 6, 12 months of follow-up
  The following biomarker analyses are implemented in the trial:
  * ELISpot/CTLp
  * EBV/CMV/BKV load + CMV/EBV T-Ly
  * Multi-parameter flow cytometry
  * gene expression profiling
  * alloantibodies
  * urinary IP-10
  * HO-1 polymorphisms
  * histology (protocol/induced biopsies)
Incidence of death by 12 months post-transplantation | 12 months post-transplantation
  incidence of death by 12 month post transplantation
Incidence of graft loss by 12 months post-transplantation | 12 months post-transplantation
  Incidence of graft loss by 12 months post-transplantation
Incidence of metabolic and cardiovascular co-morbidity by 12 months post-transplantation | 12 months post-transplantation
  Incidence of metabolic and cardiovascular co-morbidity by 12 months post-transplantation (post-transplant diabetes mellitus, dyslipidemia, hypertension, myocardial infarction, stroke, peripheral vascular disease)
Proportion of subjects who remain on tacrolimus/steroids therapy at 12 months post-transplantation | 12 months post-transplantation
  Proportion of subjects who remain on tacrolimus/steroids therapy at 12 months post-transplantation
Incidence of acute and chronic lesions assessed by the Banff 07 score in protocol biopsy at 12months post-transplantation | 12 months post-transplantation
  Banff classification:
  * Normal
  * Antibody mediated rejection
  * Borderline
  * T cell mediated rejection:
  Type IA: cases with significant interstitial infiltration (> 25% of parenchyma affected, i2 or i3) & foci of moderate tubulitis (t2) Type IB: cases with significant interstitial infiltration (> 25% of parenchyma affected, i2 or i3) & foci of severe tubulitis (t3) Type IIA: cases with mild to moderate intimal arteritis (v1) Type IIB: cases with severe intimal arteritis comprising > 25% of luminal area (v2) Type III: cases with transmural arteritis or arterial fibrinoid change & necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation (v3) Chronic allograft arteriopathy
  - Interstitial fibrosis and tubular atrophy: Grade I: mild interstitial fibrosis & tubular atrophy Grade II: moderate interstitial fibrosis & tubular atrophy Grade III: severe interstitial fibrosis & tubular atrophy/loss
Incidence of discontinuation of study treatment | 12 month
  Incidence of discontinuation of study treatment
Donor specific antibody (DSA) at 12M | 12 months post-transplantation
  Assessment of donor specific antibody at 12M Method of assessment: Luminex assay
Overall safety of tacrolimus/steroids therapy immunosuppressive regimen measured by the occurrence of viral and bacterial infections, malignancies and autoimmunity. | 12 month
  Overall safety of tacrolimus/steroids therapy immunosuppressive regimen measured by the occurrence of viral and bacterial infections, malignancies and autoimmunity
Health-related quality of life using SF-36v2 questionnaires at baseline (pre Transplantation), Month 1, Month 3, Month 6, and Month 12 | baseline (pre transplantation), Month 1, Month 3, Month 6, and Month12
  The SF-36v2 provides scores for each of the eight health domains and psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health
Assessment of patient-specific resource consumption using a trial specific questionnaire at initial discharge, Month 3, Month 6, Month 12, and in cases of repeated hospitalization | initial discharge, Month 3, Month 6, Month 12, and in cases of repeated hospitalization
  The questionnaires capture relevant apsects of resource consumption:
  * In which ward(s) a patient was hospitalized
  * Additional services (diagnostics / procedures / operations)
  * Potential dialysis procedures (past and expected frequency in the future)
  * Potential outpatient visits and the services consumed
  * Employment status and potential depency on care-giving The completion requires a review of inpatient records. Part II and Part III also require a short interview with the patient about potential outpatient visits during the study period, their employment status, and potential depedency on care-giving.
Health-related quality of life using EQ5D-5L questionnaires at baseline (pre Transplantation), Month 1, Month 3, Month 6, and Month 12 | baseline (pre transplantation), Month 1, Month 3, Month 6, and Month12
  EQ-5D is a standardized instrument for measuring generic health status. It has been widely used in population health surveys, clinical studies, economic evaluation and in routine outcome measurement in the delivery of operational healthcare.
  The EQ-5D-5L is a Patient Reported Outcome (PRO) instrument that can generally assess the quality of life of patients, regardless of their disease, over 6 questions. It also includes a vertical EQ visual analog scale (EQ VAS, 0-100 points) and a descriptive EQ-5D-5L system, which considers the following 5 dimensions or subscales over 5 levels or possible answers.
  dimensions: mobility, self-sufficiency, General Activities, Pain / Physical complaints, fear / dejectedness levels: Level 1: No problems/ No pain/ Not afraid; Level 2: Slight problems/ Slight pain/ A little anxious; Level 3: Moderate problems/ Moderate pain/ Moderate anxiety; Level 4: Major problems / Severe pain/ Very anxious; Level 5: Not able to/ Extreme pain/ Extremely anxious

CONTACTS AND LOCATIONS:
Overall Officials: Reinke Reinke, PhD, MD, Study Chair — Charité-University Medicine (Berlin, Germany); Ondrej Viklicky, PhD, MD, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Charité University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Viklicky O, Zahradka I, Bold G, Bestard O, Hruba P, Otto NM, Stein M, Sefrin A, Modos I, Meneghini M, Crespo E, Grinyo J, Volk HD, Christakoudi S, Reinke P. Tacrolimus After rATG and Infliximab Induction Immunosuppression-RIMINI Trial. Transplantation. 2024 Jan 1;108(1):242-251. doi: 10.1097/TP.0000000000004736. Epub 2023 Aug 1. PMID 37525369